CLINICAL TRIAL: NCT04079751
Title: Radiostereometric Analysis (RSA) of the ATTUNE Knee System: A Randomized Controlled Trial Comparing Anatomic (Femur First) to Neutral Mechanical Alignment Techniques
Brief Title: Trial Comparing Alignment Techniques - RSA of ATTUNE Knee System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2018-139
Record Dates: First submitted 2019-07-17; First posted 2019-09-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either Neutral mechanical alignment or Anatomical alignment using randomly generated numbers permuted in blocks of 4.
Who Masked: Participant
Masking Description: The patient will not be informed of their study allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Neutral Mechanical Alignment (Active Comparator): Total knee arthroplasty: Neutral Mechanical Alignment vs Anatomical Alignment
  Interventions: Procedure: Neutral Mechanical Alignment
- Anatomical Alignment (Active Comparator): Total knee arthroplasty: Neutral Mechanical Alignment vs Anatomical Alignment
  Interventions: Procedure: Anatomical Alignment

INTERVENTIONS:
Procedure: Neutral Mechanical Alignment — Hip-knee-ankle angle of 180° ± 3°.
  Arms: Neutral Mechanical Alignment
Procedure: Anatomical Alignment — Restoring a patient's pre-diseased limb alignment
  Arms: Anatomical Alignment

SUMMARY:
The purpose of this study is to compare migration patterns between mechanical and anatomic alignment surgical techniques for the Attune S+ CR-FB knee system using model-based RSA over the first 2 post-operative years.

DETAILED DESCRIPTION:
This is a multi-centre, randomized controlled trial of patients undergoing cruciate-retaining total knee arthroplasty with the Attune S+ fixed bearing TKR system. Patients will be randomized to two study groups:

1. Neutral mechanical alignment;
2. Anatomical alignment.

The principal objective of this study is to compare migration patterns between mechanical and anatomic alignment surgical techniques for the Attune S+ CR-FB knee system using model-based RSA over the first 2 post-operative years.

Secondary objectives include; comparison of 2-year migration values against published thresholds for adequate short-term fixation, comparison of functional and health status of subjects following surgery, comparison of intra-operative soft-tissue releases, incidence of complications and adverse events, and to assess several health economic parameters relating to the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic osteoarthritis of the knee indicating primary total knee arthroplasty
2. Varus knee deformity of 0 to 10 degrees
3. Sufficient ligamentous function to warrant retention of the posterior cruciate ligament
4. Between the ages of 21 and 80 inclusive
5. Patients willing and able to comply with follow-up requirements and self-evaluations
6. Ability to give informed consent

Exclusion Criteria:

1. Active or prior infection
2. Medical condition precluding major surgery
3. Inflammatory arthropathy
4. Prior patellectomy
5. PCL deficiency
6. Major Coronal plane deformity
7. Valgus alignment
8. Bone defects requiring augments, cones and/or stemmed implants
9. Body Mass Index 45 or more

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Implant migration | 2 years
  Measured via radiosteriometric analysis (RSA)

SECONDARY OUTCOMES:
Oxford-12 knee score | Pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years
  The Oxford Knee Score (OKS) is a patient self-administered 12-item questionnaire with each question having a Likaert-like response option. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance. The OKS measures pain and general activities of daily living.
Pain Catastrophizing Scale (PCS) | Pre-operative, 12 months
  The patient are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain. Each PCS item is rated on a 5-point scale: 0 (not at all) to 4 (all the time). The PCS total score is computed by summing responses to the 13 items. PCS total scores range from 0 - 52.
European Quality of Life (EQ-5D-5L) | Pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in functional outcomes assessments. The EuroQol 5D 5L questionnaire is a standardized instrument for use as a measure of generic health status - completed by the subject. The EQ5D uses a Likert scale which assesses five states (mobility, self care, usual care, pain and discomfort and anxiety and depression) at five different levels - none(0), slight(1), moderate(2), severe(3) or unable to perform(5). Levels are coded 1-5 and an index score is then generated.
Pre-operative Patient's Knee Implant Performance (PKIP) | Pre-operative, 6 weeks, 3 months, 6 months, 1 year, 2 years
  The Pre-surgical and/or Post-surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient reported questionnaire that consists of 24 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likaert- like response option.
7. University of California at Los Angeles (UCLA) Activity Level scale | Pre-operative, 6 months, 1 year, 2 years
  Evaluate and compare the change in UCLA activity score compared to baseline in the study cohort. UCLA activity scores range from 1 to 10, and is a measure of activity with 10 being most active.
Pain VAS | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year, 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported satisfaction as measured using the visual analogue scale (VAS) from 0 (No pain) - 100 (Worst pain imaginable)
Patient satisfaction: VAS | Preoperative, 3 Months, 6 Months, 1 Year, 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported pain severity as measured using the visual analogue scale (VAS) from 0 (Unsatisfied) - 100 (Completely satisfied)
Patient complications | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year, 2 Years
  Evaluate the type and frequency of the complications/adverse events.
Hospital stay | Up to 1 week
  Number of days in hospital
Tourniquet time | Intraoperative
  Length of time tourniquet was applied (minutes)
Length of surgery | Intraoperative
  Length of surgery, from open to closing of incision (minutes)
Blood loss | Intraoperative
  Amount of blood loss during the procedure (mL)
Anesthesia type | Intraoperative
  Anesthesia methods (general, spinal, epidural, TXA)
Peri-operative pain management | Intraoperative
  A tabulation of the pain management (Peri-Articular Injection, Femoral Nerve Block, Add. Canal Block or none) used during the procedure.
Soft tissue release | Intraoperative
  A tabulation of the tissue released during the procedure (MCL, LCL, PCL, Posterior Capsule Release).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, Principal Investigator — Concordia Joint Replacement Group
Locations (2):
- Canada (2):
  - Concordia Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario